CLINICAL TRIAL: NCT03791021
Title: Developing a Postpartum Depression Predicting Tool, During the Third Trimester of Pregnancy
Brief Title: Early Diagnosis of PPD Through Self-portraits
Acronym: ppd
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: University of Haifa (Other)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Other Study IDs: 5651-18-SMC
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Postpartum Depression
Keywords: postpartum, depression, self portraits
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- third trimester pregnant women: the group of participants in this research would include approximately 100 subjects in the third trimester of their pregnancy. the participants would be collected in the central area of Israel from various socioeconomic groups. each participant would be asked to make draw a person (DAP) test, and answer a number of questionnaires including Edinburgh Postnatal Depression Scale (EPDS), Beck Depression Inventory II (BDI-II), and Traumatic Events Questionnaire (TEQ).
  Interventions: Diagnostic Test: draw a person (DAP); Diagnostic Test: Edinburgh Postnatal Depression Scale (EPDS); Diagnostic Test: Beck Depression Inventory- II (BDI-II); Diagnostic Test: Traumatic Events Questionnaire (TEQ)

INTERVENTIONS:
Diagnostic Test: draw a person (DAP) — the subjects will be given a blank sheet of white paper and a pencil, and will be asked to draw themselves with no other additional instructions.
Diagnostic Test: Edinburgh Postnatal Depression Scale (EPDS) — measure of postpartum depression symptoms.
Diagnostic Test: Beck Depression Inventory- II (BDI-II) — BDI-II is based on clinical observations of behaviors associated with depression, and it retains the somatic items in accordance with the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria related to loss of energy. ansd sleep disturbances.
Diagnostic Test: Traumatic Events Questionnaire (TEQ) — The TEQ assesses experiences with nine specific types of traumatic events (e.g., accidents, crime, adult abusive experiences) reported in the empirical literature as having the potential to elicit PTSD symptoms.

SUMMARY:
the target of the research is development of a predictive tool for early identification of women which are at higher risk for development of postpartum depression.

the evaluating tools include self portraits and questionnaire during the third trimester of pregnancy.

The suggested research aims to evaluate if and how it would be possible to predict the potential for postpartum mood swing disorders in pregnant women while in the third trimester. The later to prevent the mother from enduring such a detrimental experience, which influences the child development, the family as well as the mother's intimate relationship.

The aim is to identify indicators to predict such potential, using questionnaires and self-portraits during pregnancy, to allow early intervention and treatment. Early diagnosis and quick treatment of pregnant women or post-partum mothers will allow them a higher level of functioning and may even prevent eventually infant neurological and developmental delays and hardships.

DETAILED DESCRIPTION:
the target of the research is to evaluate a method based on self portraits and targeted questionnaire done in the third trimester and three months later in order to identify pregnant women in higher risk to develop PPD.

the minimal number of objectives participating in the research would be 100 pregnant women during the third trimester of pregnancy.

the Draw A Person (DAP) test was described by Machover in 1949. it is still considered a reliable and well recognized test for evaluation of mental stress and disorders (Gilory, 2012).

in the research approximately 100 pregnant women in the third trimester would be asked to draw a self portrait in two different time points (during the third trimester and three to six months postpartum). in addition to the self portraits the participants would be asked to fill a set of questionnaires to evaluate the degree of depression, self esteem, personal history of traumatic events, and demographic data.

the self portraits would be evaluated by three judges. the reliability between judges would be tested using KAPPA test.

ELIGIBILITY:
Inclusion Criteria:

* third trimester pregnant women

Exclusion Criteria:

* pregnant women with established diagnosis of mental disorders
* still birth or intra uterine disorders

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 100 pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
development of a reliable projective tool for prediction of PPD | one year
  ratification of a projective tool using self portrait tests to identify patient at risk for developing PPD

CONTACTS AND LOCATIONS:
Locations (1):
- Aya Mohr Sasson, Ramat Gan, Please Select, Israel